CLINICAL TRIAL: NCT01868360
Title: Subconjunctival Aflibercept Injection for Corneal Neovascularization
Brief Title: Using Aflibercept Injection to Treat Blood Vessel Growth Over the Cornea
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Balamurali Ambati (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Balamurali Ambati, Professor of Ophthalmology, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMB65110
Record Dates: First submitted 2013-05-15; First posted 2013-06-04 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Corneal Neovascularization
Keywords: cornea; transplant; graft; neovascularization
MeSH Terms: conditions — Corneal Neovascularization; Corneal Diseases; Neovascularization, Pathologic | interventions — aflibercept; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A subconjunctival aflibercept (Experimental): Patients will receive 2mg (0.05mL) subconjunctival aflibercept injection in addition to standard of care treatment (steroids and cyclosporine). Patients will receive one injection four weeks (+/- 1 week) prior to transplantation. They will receive a second injection at the conclusion of corneal transplantation.
  Patients may receive as-needed repeat injections (minimum of 30 days in between treatments) for recurrence of corneal neovascularization (defined as >1.0 mm crossing onto the cornea, past the limbus, or extension of vessels beyond previously documented extent) during the follow-up period.
  Interventions: Drug: Subconjunctival aflibercept
- Group B: Standard of care only (Placebo Comparator): Patients will receive standard of care (steroids and cyclosporine) treatment only.
  Interventions: Other: Placebo: Standard of care only

INTERVENTIONS:
Drug: Subconjunctival aflibercept — subconjunctival aflibercept injection
  Other Names: EYLEA®; VEGF Trap-Eye
  Arms: Group A subconjunctival aflibercept
Other: Placebo: Standard of care only — Patients will receive standard of care (steroids and cyclosporine) treatment only.
  Other Names: Standard of care
  Arms: Group B: Standard of care only

SUMMARY:
The cornea is the clear front part of the eye. Corneal neovascularization, the excessive growth of blood vessels into the cornea, is a sight-threatening condition. Corneal neovascularization is also a well recognized risk factor for corneal graft failure. The current standard of care to prevent graft rejection includes use of topical steroids and medicines that suppress the immune system. These medicines do not address corneal neovascularization. The purpose of the study is to establish the safety and potential efficacy of subconjunctival injections of aflibercept (EYLEA® , marketed by Regeneron) injection in inducing regression of blood vessels growing into the cornea and promoting graft survival.

This study is being conducted by Dr. Balamurali Ambati at the Moran Eye Center.

DETAILED DESCRIPTION:
Corneal neovascularization is a sight threatening condition and is also a well recognized risk factor for corneal graft failure. Current standard of care to prevent graft rejection includes use of topical steroids and immunosuppressants. These do not address corneal neovascularization. The cornea is kept in its avascular state by a complex interaction of signal proteins and host receptors, with a vital role played by the soluble VEGF-receptor 1. In any condition of chronic corneal inflammation or hypoxia, the balance may tip in favour of pro-angiogenic factors, and neovascularization will ensue. Early and limited studies have examined the effect of subconjunctival or intracorneal administration of monoclonal antibodies to VEGF (bevacizumab, ranibizumab) in combating corneal neovascularization. Most report subtotal or temporary regression. The development of aflibercept (also known as VEGF Trap-Eye) offers new hope of more effectively combating the problem. In this study, research will be conducted to investigate and assess safety of subconjunctival aflibercept injection in patients with corneal neovascularization undergoing corneal transplantation.

This is a phase 1, prospective, randomized, open label clinical trial that will enroll 10 corneal transplant patients with corneal neovascularization in one or more quadrants crossing more than 0.5 mm over the limbus at the time of corneal transplantation.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet the following criteria to be eligible for inclusion in the study:

1. Candidates for corneal transplantation (only one eye per patient would be enrolled)
2. Patients with corneal neovascularization in one or more quadrants crossing more than 1.0 mm over the limbus at time of enrollment in the study
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent
5. Age 18 or over

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

1. Patients receiving antiangiogenic anti-VEGF medication either systemically or intravitreally for other pathology or have received these drugs within 3 months of study enrollment
2. Patients with active corneal infection requiring additional treatment modalities
3. Patients receiving coumadin with INR >2.0, other anti-thrombotic agents (e.g., aspirin, Plavix) permitted at discretion of investigator
4. History of cerebrovascular accident or myocardial infarction within 6 months prior to study enrollment
5. Uncontrolled blood pressure- defined as SBP>160 mmHg or DBP >95mmHg while patient is sitting
6. Pregnant or breast-feeding women
7. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly) *Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety defined by incidence and severity of adverse events at week 28 | Week 28
  The primary endpoint in the study is safety as defined by incidence and severity of adverse events in patients with corneal neovascularization undergoing corneal transplant.

SECONDARY OUTCOMES:
neovascularization regression | at time of transplant
  Ability of subconjunctival aflibercept injection to regress neovascularization at time of transplant and promote graft survival after corneal transplantation
Need for immunosuppression | Week 28
  Need for immunosuppression at week 28 in both treatment groups
Effect on corneal infections | Through week 28
  Effect on corneal infections or other side effects through week 28 in both treatment groups
Change in visual acuity | Week 28
  Change in ETDRS visual acuity from baseline at week 28 in both treatment groups
Mean number of injections | Week 28
  Mean number of injections performed per patient through week 28 in patients receiving subconjunctival aflibercept injections
Rescue therapy | Week 28
  Need for rescue treatment in the standard of care group through week 28
neovascularization regression | at 28 weeks after transplant
  Ability of subconjunctival aflibercept injection to regress neovascularization (at 28 weeks after transplant) and promote graft survival after corneal transplantation
neovascularization regression | at 52 weeks after transplantation
  Ability of subconjunctival aflibercept injection to regress neovascularization at 52 weeks after transplant and promote graft survival after corneal transplantation
Need for immunosuppression | week 52
  need for immunosuppression at week 52 in both treatment groups
Effect on corneal infections | Through week 52
  Effect on corneal infections or other side effects through week 52 in both treatment groups.
Change in visual acuity | Week 52
  Change in ETDRS visual acuity from baseline at week 52 in both treatment groups
Mean number of injections | Week 52
  Mean number of injections performed per patient through week 52 in patients receiving subconjunctival aflibercept injections
Rescue therapy | Week 52
  Need for rescue treatment in the standard of care group through week 52

CONTACTS AND LOCATIONS:
Overall Officials: Balamurali Ambati, M.D., Ph.D., M.B.A., Principal Investigator — University of Utah
Locations (1):
- John A. Moran Eye Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] The collaborative corneal transplantation studies (CCTS). Effectiveness of histocompatibility matching in high-risk corneal transplantation. The Collaborative Corneal Transplantation Studies Research Group. Arch Ophthalmol. 1992 Oct;110(10):1392-403. PMID 1417537
- [Background] Chang JH, Garg NK, Lunde E, Han KY, Jain S, Azar DT. Corneal neovascularization: an anti-VEGF therapy review. Surv Ophthalmol. 2012 Sep;57(5):415-29. doi: 10.1016/j.survophthal.2012.01.007. PMID 22898649
- [Background] Chang JH, Gabison EE, Kato T, Azar DT. Corneal neovascularization. Curr Opin Ophthalmol. 2001 Aug;12(4):242-9. doi: 10.1097/00055735-200108000-00002. PMID 11507336